CLINICAL TRIAL: NCT03314792
Title: A Comparison of Analgesic and Respiratory Effects From Tapentadol Versus Oxycodone After Laparoscopic Hysterectomy.
Brief Title: Effects of Tapentadol Versus Oxycodone After Hysterectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Harald Lenz, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/776
Record Dates: First submitted 2017-09-25; First posted 2017-10-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative; Pain Uterus; Pain, Acute; Opioid Use; Analgesics, Antipyretics, and Antirheumatics Causing Adverse Effects in Therapeutic Use; Visceral Pain
Keywords: pain; postoperative pain; postoperative pain management; opioid; analgesia; oxycodone; tapentadol; hysterectomy; respiratory depression
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Visceral Pain; Pain; Agnosia; Respiratory Insufficiency | interventions — Tapentadol; Oxycodone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients were not told which medicine they were given, but due to difference in apperance of pills they would be able to find out which medicine they were given if they wanted to. Care providers at the hospital ward administering the medication would know which medicine were given due to apperance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone (Active Comparator): Active comparator drug administrated.
  Interventions: Drug: Oxycodone
- Tapentadol (Experimental): Experimental drug administrated.
  Interventions: Drug: Tapentadol

INTERVENTIONS:
Drug: Tapentadol — * Palexia depot 50 mg® (tapentadol depot 50 mg): Administered by the patient as oral premedication 1 hour before scheduled start of surgery. Palexia depot is repeated once after 12 hours.
  * Palexia 50 mg® (tapentadol 50 mg): Administered as oral rescue medicine. First possible administration in postoperative ward when the patient is awake and available for oral medication. Maximum 4 tablets/24-hour study period. Minimum 1 hour 15 minutes between tablets. The patient is instructed to take 1 tablet if pain is increasing and the minimum period since last tablet is exceeded.
  Arms: Tapentadol
Drug: Oxycodone — * OxyContin 10 mg® (oxycodone extended-release 10 mg): Administered by the patient as oral premedication 1 hour before scheduled start of surgery. OxyContin is repeated once after 12 hours.
  * OxyNorm 10 mg® (oxycodone immediate-release 10 mg): Administered as oral rescue medicine. First possible administration in postoperative ward when the patient is awake and available for oral medication. Maximum 4 capsules/24-hour study period. Minimum 1 hour 15 minutes between capsules. The patient is instructed to take 1 tablet if pain is increasing and the minimum period since last tablet is exceeded.
  Arms: Oxycodone

SUMMARY:
Opioids remain the first-line drugs for the treatment of moderate to severe postoperative pain, but the use is limited by well-known side-effects, most of which are dose-dependent.

The opioid oxycodone is standard therapeutic treatment for acute postoperative pain, either in immediate-release formulation, OxyNorm®, or as extended-release formulation, OxyContin®. Oxycodone provides analgesic effects through µ-opioid receptors in the central nervous system.

Tapentadol hydrochloride/depot (Palexia/depot®) is a novel, centrally acting, strong analgesic with a dual mechanism of action on µ-opioid receptors and noradrenaline reuptake in the central nervous system. Tapentadol is an active compound, devoid of active metabolites and not reliant on enzyme systems. For these reasons, it has a low drug interaction potential. This dual mechanism also translates clinically into less adverse effects than with pure opioid agonists like oxycodone. This is probably due to less µ-opioid receptor stimulation.

Tapentadol has been shown effective in models of acute, osteoarthritic, neuropathic and cancer pain. There is now an increasing use of tapentadol in postoperative pain treatment in Norway. However, there is a lack of broad-based evidence for the use of tapentadol in the post-surgical setting. So far, to our knowledge, there are only published studies on postoperative pain treatment after orthopedic and dental surgery, but none related to deep abdominal pain.

Tapentadol is shown in several studies on chronic pain patients to have comparable analgesic effects to traditional opioid pain medications like oxycodone and morphine, but with a more tolerable side-effect profile. In the postoperative setting after dental or orthopedic surgery, studies have shown less nausea and constipation. It has also been suggested a lower frequency of pruritus compared with oxycodone, but no difference in central nervous system symptoms such as sleepiness or dizziness. The most dangerous side-effect from opioids is respiratory depression with the potential of fatal outcome. The investigators have not found any publications from short-term postoperative pain management comparing the respiratory effect of tapentadol to the traditional opioids.

The aim of the study is to compare the analgesic effect and side-effects of this new analgesic, tapentadol, to the standard treatment to day, oxycodone, in the acute postoperative period after hysterectomy.

DETAILED DESCRIPTION:
Postoperative pain is a major cause of postoperative suffering, prolonged hospitalization, complications and increased costs. It has been shown that postoperative pain is a frequent and unresolved problem in Norwegian hospitals, and so also internationally. Building knowledge on pain prophylaxis and treatment of postoperative pain is an area with substantial potential for improvement and affecting many patients.

Opioids remain as first-line drugs for the treatment of moderate to severe postoperative pain, but the use is limited by well-known side-effects, most of which are dose-dependent.

The opioid oxycodone is used as standard therapeutic treatment for acute postoperative pain, either in immediate-release formulation, OxyNorm®, or as extended-release formulation, OxyContin®. Oxycodone is a pure opioid receptor agonist with central and peripheral effects.

Tapentadol hydrochloride/depot (Palexia/depot®) is a novel, centrally acting, strong analgesic with a dual mechanism of action. It is a µ-opioid receptor agonist with central and peripheral effects, and it also inhibits noradrenaline reuptake in the central nervous system. Tapentadol is an active compound, devoid of active metabolites and not reliant on enzyme systems. For these reasons, it has a low drug interaction potential.

Opioid receptors are usually not well expressed in non-inflamed peripheral tissue and they have limited effect on the peripheral pathophysiology and origin of acute wound pain. While postoperative pain basically is induced by relevant nociceptive pain nerve stimulation, there is also a neuropathic component in most cases. Opioids are not very effective in blocking neuropathic pain in low to moderate doses. Also, opioids do not have the potential to block the wind-up of pain when given before the start of surgical trauma. The noradrenaline re-uptake inhibition (NRI) component of tapentadol is believed to have effect on descending pathways in the spinal cord. Such excitatory and inhibitory pathways act through monoamine systems mediated by noradrenaline and 5-hydroxytryptamine (5-HT). The inhibition of noradrenaline reuptake increases monoaminergic transmission in the descending pain inhibitory pathways, leading to reduced pain sensation. It seems like tapentadol produce not simply additive, but synergistic anti-nociceptive action by inhibitory actions in µ-opioid receptor agonism and NRI. While the effect on µ-opioid receptors is important in nociceptive pain, the NRI component seems to be especially relevant for both acute and persistent neuropathic pain.

Tapentadol has been shown effective in models of acute, osteoarthritic, neuropathic and cancer-induced bone pain. There is now an increasing use of tapentadol in postoperative pain treatment in Norwegian hospitals. However, there is a lack of broad-based evidence for the use of tapentadol in the post-surgical setting. So far, to our study group's knowledge, there are only published studies on postoperative pain treatment after orthopedic and dental surgery, but none related to visceral pain. Most studies have so far been initiated by the industry. The standard treatment today, oxycodone, on the other hand is shown in several studies to have a preferable analgesic effect on pain of visceral origin compared to morphine.

The synergistic effect of µ-opioid receptor agonism and NRI translates clinically into less adverse effects than with pure opioid agonists. This is probably due to less µ-opioid receptor stimulation. Tapentadol is shown in several studies on chronic pain patients to have comparable analgesic effects to traditional opioid pain medications like oxycodone and morphine, but with a more tolerable side-effect profile. In the postoperative setting after dental or orthopedic surgery, studies have shown less nausea and constipation. It has also been suggested a lower frequency of pruritus compared with oxycodone, but no difference in central nervous system symptoms such as somnolence or dizziness. The most dangerous side-effect from opioids is respiratory depression with the potential of fatal outcome. Intravenous oxycodone is shown to have dose dependent effect on respiratory depression decreasing the mean minute volume with a more rapid onset than morphine. One study has attempted to study respiratory depression after tapentadol administration, but failed due to technical failure of the pulse oximetry device. The investigators have not found any other publications from short-term postoperative pain management comparing any respiratory effect of tapentadol to the traditional opioids.

The aim of the study is to compare the analgesic effect and side-effects of this new analgesic, tapentadol, to the standard treatment to day, oxycodone, in the acute postoperative period in patients with visceral pain. Patients scheduled for elective hysterectomy are chosen as the study population, as this is a group of patients with significant visceral pain after surgery.

The study will be performed as a randomized, double-blind, prospective, parallel-group, single-center study on patients scheduled for laparoscopic sub-/total hysterectomy, as this is a classic study comparing effects from two different medications on two groups in a population.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with a benign gynecological condition, undergoing laparoscopic, supra-cervical or total hysterectomy in general anesthesia.
* Age 18-64 years.
* ASA (American Society of Anesthesiologists) classification I-III.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Conference on Harmonisation GCP, and national/local regulations.
* The patients will be recruited from the patient population at the Department of Gynaecology.

Exclusion Criteria:

* Age under 18 or over 65.
* BMI > 31 and/or weight <55 kg, >85 kg.
* Chronic pain syndromes related to organ systems other than the female reproductive system.
* Chronic opioid therapy (codeine medication allowed up to 60 mg/day) or enteral steroid therapy.
* Alcohol or medical abuse/addiction.
* Chronic obstructive pulmonary disease (spirometry with postbronchodilator FEV1/FVC ratio less than 0.7), untreated asthma (FEV1/FVC is reduced to less than 0.70), obstructive sleep apnea or other conditions known to predispose for respiratory depression.
* Neurological diagnosis with affection of respiratory system or prone to seizures.
* Previously diagnosed kidney (glomerular filtration rate <60 mL/min/1.73 m2 over 3 months) or liver impairment (ALAT > 45 U/L; ASAT > 35 U/L; ALP > 105 U/L; GT > 45 U/L age 18-39 or GT > 75 U/L age over 39; LD > 205 U/L).
* Biliary tract disease.
* Paralytic ileus.
* Heart failure (NYHA III-IV).
* Malignancy of any kind under treatment. Malignancy during last 5 years.
* HIV infection. Infections of any kind affecting the patient's clinical status, i.e. upper or lower airway infection, urinary tract infection, deep wound infection. Infections not affecting the patient's clinical status, i.e. conjunctivitis, is not an exclusion criteria.
* Untreated depression, severe anxiety or other psychiatric disorders independent of treatment.
* Nursing mothers.
* Cognitive failure, language barriers, hearing/visual disability or other factors which make follow-up difficult.
* Allergy or contraindication to any of the medications used in the study.
* Lactose intolerance.
* Monoamine oxidase inhibitors or SNRI (serotonin norepinephrine reuptake inhibitors) within 14 days prior to randomization. SSRI (selective serotonin reuptake inhibitors) use is not an exclusion criterion if stable dose for at least 30 days before screening.
* H1-antihistamine is not an exclusion criterion unless the patient experiences somnolence as a side-effect.
* The concurrent use of benzodiazepines, barbiturates, neuroleptics, phenytoin tricyclic antidepressants, gabapentinoids, tramadol, clonidine, cimetidine, rifampicin, protease inhibitors, St John's wort (Hypericum perforatum), macrolides and antimycotics such as ketoconazole and fluconazole is not allowed.
* Known complications to anesthesia or difficult airway (Definition of difficult airway: "The clinical situation in which a conventionally trained anesthesiologist experiences difficulty with mask ventilation, difficulty with tracheal intubation, or both.").
* Patients who have participated in other clinical trials during the last 6 months are excluded to avoid confounders to the current study and for patient safety reasons.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Pain 1 hour postoperatively. | 1 hour
  Difference in scoring of pain at rest using the numerical rating scale for pain between the two intervention groups, tapentadol and oxycodone.

SECONDARY OUTCOMES:
Pain 2 hours postoperatively. | 2 hours
  Difference in scoring of pain at rest using the numerical rating scale for pain between the two intervention groups, tapentadol and oxycodone.
Pain 3 hours postoperatively. | 3 hours
  Difference in scoring of pain at rest using the numerical rating scale for pain between the two intervention groups, tapentadol and oxycodone.
Pain 24 hours postoperatively. | 24 hours
  Difference in scoring of pain at rest using the numerical rating scale for pain between the two intervention groups, tapentadol and oxycodone.
Pain relief 30 minutes | 30 minutes
  Pain relief, measured with categorical scale "none, slight, moderate, good or complete", comparing pain at 30 minutes postoperatively to the previous measurement point. The measure "total pain relief" (TOTPAR) will be calculated from these values.
Pain relief 1 hour | 1 hours
  Pain relief, measured with categorical scale "none, slight, moderate, good or complete", comparing pain at 1 hour postoperatively to the previous measurement point. The measure "total pain relief" (TOTPAR) will be calculated from these values.
Pain relief 2 hours | 2 hours
  Pain relief, measured with categorical scale "none, slight, moderate, good or complete", comparing pain at 2 hours postoperatively to the previous measurement point. The measure "total pain relief" (TOTPAR) will be calculated from these values.
Pain relief 3 hours | 3 hours
  Pain relief, measured with categorical scale "none, slight, moderate, good or complete", comparing pain at 3 hours postoperatively to the previous measurement point. The measure "total pain relief" (TOTPAR) will be calculated from these values.
Pain relief 24 hours | 24 hours
  Pain relief, measured with categorical scale "none, slight, moderate, good or complete", comparing pain at 24 hours postoperatively to the previous measurement point. The measure "total pain relief" (TOTPAR) will be calculated from these values.
Global medication performance | 24 hours
  The measure "Global medication performance" after 24 hours: the patient evaluates the overall satisfaction with the pain treatment on a scale ("poor, fair, good, very good, excellent").
Time to first rescue medicine | 24 hours
  Time to first intravenous and/or per oral rescue medicine.
Total rescue analgesic consumption | 24 hours
  Total intravenous and per oral rescue analgesic consumption over 24 hours.
Respiratory depression | 24 hours
  Continuous measurement of end-tidal carbon dioxide (ETCO2) with Smart CapnoLine® Plus (Microstream®), data are collected at postoperatively.
Respiratory rate | 24 hours
  Respiratory rate at rest is measured postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Lenz, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The study has no collaborators outside Oslo University Hospital and individual participant data (IPD) is not planned shared with other researchers during the study periode. The database with IPD will be stored in a secure research server at Oslo University Hospital according to the policy for secure storage.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The database will be stored until 31.12.2035.
Access Criteria: Sponsor's representatives (e.g. monitors, auditors) and/or competent authorities will be allowed access to source data for source data verification.
  The sponsor has the right to share IPD underlying the results presented in the final published article should any journal or editor require this. The data underlying the results are defined as the IPD required to reproduce the article's findings, including necessary metadata.
  Other research groups may be granted access to the data upon request after publishing of the article. This will be according to the relevant journal's requirements for data sharing upon publishing. The research must have relevant connection to the original study and the research group must fulfill requirements for safe storage and handling of data. The patients are informed of potential data sharing in the informed consent form. The confidentiality guidelines of Oslo University Hospital and the regional ethics committee will at all times be followed.

REFERENCES:
- [Background] Langford RM, Knaggs R, Farquhar-Smith P, Dickenson AH. Is tapentadol different from classical opioids? A review of the evidence. Br J Pain. 2016 Nov;10(4):217-221. doi: 10.1177/2049463716657363. Epub 2016 Jul 25. PMID 27867511
- [Background] Raeder J. Opioids in the treatment of postoperative pain: old drugs with new options? Expert Opin Pharmacother. 2014 Mar;15(4):449-52. doi: 10.1517/14656566.2014.879292. Epub 2014 Jan 17. PMID 24437530
- [Background] Schroder W, Vry JD, Tzschentke TM, Jahnel U, Christoph T. Differential contribution of opioid and noradrenergic mechanisms of tapentadol in rat models of nociceptive and neuropathic pain. Eur J Pain. 2010 Sep;14(8):814-21. doi: 10.1016/j.ejpain.2010.05.005. Epub 2010 Jun 11. PMID 20541444
- [Background] Riley J, Eisenberg E, Muller-Schwefe G, Drewes AM, Arendt-Nielsen L. Oxycodone: a review of its use in the management of pain. Curr Med Res Opin. 2008 Jan;24(1):175-92. doi: 10.1185/030079908x253708. PMID 18039433
- [Background] Kleinert R, Lange C, Steup A, Black P, Goldberg J, Desjardins P. Single dose analgesic efficacy of tapentadol in postsurgical dental pain: the results of a randomized, double-blind, placebo-controlled study. Anesth Analg. 2008 Dec;107(6):2048-55. doi: 10.1213/ane.0b013e31818881ca. PMID 19020157
- [Background] Stegmann JU, Weber H, Steup A, Okamoto A, Upmalis D, Daniels S. The efficacy and tolerability of multiple-dose tapentadol immediate release for the relief of acute pain following orthopedic (bunionectomy) surgery. Curr Med Res Opin. 2008 Nov;24(11):3185-96. doi: 10.1185/03007990802448056. Epub 2008 Oct 15. PMID 18851776
- [Background] Daniels SE, Upmalis D, Okamoto A, Lange C, Haeussler J. A randomized, double-blind, phase III study comparing multiple doses of tapentadol IR, oxycodone IR, and placebo for postoperative (bunionectomy) pain. Curr Med Res Opin. 2009 Mar;25(3):765-76. doi: 10.1185/03007990902728183. PMID 19203298
- [Background] Hale M, Upmalis D, Okamoto A, Lange C, Rauschkolb C. Tolerability of tapentadol immediate release in patients with lower back pain or osteoarthritis of the hip or knee over 90 days: a randomized, double-blind study. Curr Med Res Opin. 2009 May;25(5):1095-104. doi: 10.1185/03007990902816970. PMID 19301989
- [Background] Lee LA, Caplan RA, Stephens LS, Posner KL, Terman GW, Voepel-Lewis T, Domino KB. Postoperative opioid-induced respiratory depression: a closed claims analysis. Anesthesiology. 2015 Mar;122(3):659-65. doi: 10.1097/ALN.0000000000000564. PMID 25536092
- [Background] Chang SH, Maney KM, Phillips JP, Langford RM, Mehta V. A comparison of the respiratory effects of oxycodone versus morphine: a randomised, double-blind, placebo-controlled investigation. Anaesthesia. 2010 Oct;65(10):1007-12. doi: 10.1111/j.1365-2044.2010.06498.x. PMID 20712805
- [Background] Ramaswamy S, Chang S, Mehta V. Tapentadol--the evidence so far. Anaesthesia. 2015 May;70(5):518-22. doi: 10.1111/anae.13080. No abstract available. PMID 25866038
- [Derived] Comelon M, Raeder J, Draegni T, Lieng M, Lenz H. Tapentadol versus oxycodone analgesia and side effects after laparoscopic hysterectomy: A randomised controlled trial. Eur J Anaesthesiol. 2021 Sep 1;38(9):995-1002. doi: 10.1097/EJA.0000000000001425. PMID 33428347

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03314792/Prot_SAP_000.pdf